CLINICAL TRIAL: NCT05698069
Title: Reliability and Validity of the Turkish Version of the Pain Modulation Index
Brief Title: Turkish Version of Pain Modulation Index
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Assistant Professor, Ege University
Other Study IDs: 21-7T/44
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic pain: Patients with non-cancer pain of more than 3 months duration.
  Interventions: Diagnostic Test: Pain Modulation Index; Other: Pain Detect; Other: Central sensitization inventory

INTERVENTIONS:
Diagnostic Test: Pain Modulation Index — A 18 item questionnaire assessing patients' pain characteristics for the detection of disordered pain modulation processes.
Other: Pain Detect — A questionnaire that was validated for the assessment of neuropathic pain
Other: Central sensitization inventory — A questionnaire developed for the detection of central sensitization.

SUMMARY:
In order to assess the validity and reliability of the Turkish version of Pain Modulation Index, 125 volunteers with chronic pain were enrolled in the study. Test and re-test method was used to assess reliability and correlation analyses with Pain Detect, visual analog scale pain and central sensitization inventory scores were used to assess validity of the questionnaire. Turkish version of the Pain Modulation Index was found to be a valid and reliable tool for evaluating chronic pain.

DETAILED DESCRIPTION:
Pain Modulation Index is a questionnaire that was developed in English for the assessment of chronic pain for qualities consistent with central sensitization. The English version of the questionnaire was translated into Turkish by two physicians than back translated into English by two separate bilingual translators. Initially 10 volunteers were asked to answer this first version of the questionnaire and report any difficulties in understanding the items. Their feedback was used to give the questionnaire its final shape. For the validation stage, patients that were diagnosed as having chronic non-cancer pain with more than 3 months duration were enrolled into the study. They answered the questions twice, 15 days apart. In addition to the Turkish version of the Pain Modulation Index, on the first visit, they were also asked to answer Pain Detect and Central Sensitization Inventory. Their answers were analysed to assess the validity and reliability of the Turkish version of Pain Modulation Index.

ELIGIBILITY:
Inclusion Criteria:

* presence of chronic non-cancer pain of more than 3 months duration

Exclusion Criteria:

* Illiteracy
* Refusal to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had non-cancer pain for more than 3 months duration.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Reliability of the Turkish version of pain modulation index | 15 days
  Internal consistency was evaluated by test retest method and calculating the coefficient alpha (α) or Cronbach's coefficient, and if the Cronbach's coefficient value was greater than 0.7, it was considered as an acceptable internal consistency
Validity of the Turkish version of Pain Modulation Index | 1 day
  Index scores were analysed for their correlation with Pain Detect and Central Sensitization Inventory scores.

CONTACTS AND LOCATIONS:
Overall Officials: Simin Hepguler, Prof, Principal Investigator — Ege University Hospital
Locations (1):
- Ege University Hospital, Department of Physical and rehabilitation medicine, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Austin PD, Asghari A, Costa DSJ, Siddall PJ. The development of a novel questionnaire assessing alterations in central pain processing in people with and without chronic pain. Scand J Pain. 2020 Apr 28;20(2):407-417. doi: 10.1515/sjpain-2019-0087. PMID 31785195